CLINICAL TRIAL: NCT03143361
Title: Outcome Comparison of Different Surgical Strategies for the Management of Severe Aortic Valve Stenosis: Study Protocol of a Prospective Multicentre European Registry (E-AVR Registry)
Brief Title: Prospective European Multicenter Study on Aortic Valve Replacement: (E-AVR Registry)
Acronym: E-AVR
Status: Recruiting | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: University of Genova (Other); University Hospitals, Leicester (Other); University of Hamburg-Eppendorf (Other); San Camillo Hospital, Rome (Other); University of Turin, Italy (Other); Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Udine, Italy (Other); Hospital Clinic of Barcelona (Other); University of Lausanne Hospitals (Other); Hopital Universitaire Robert-Debre (Other); Paracelsus Medical University (Other); University of Campania Luigi Vanvitelli (Other); University of Texas, Southwestern Medical Center at Dallas (Other); Clinique Pasteur (Other); Cardiocentro Ticino (Other); Universita di Verona (Other)
Responsible Party: Principal Investigator, Francesco Onorati, MD, PhD, Associate Professor of Cardiac Surgery, Universita di Verona
Other Study IDs: E-AVR
Record Dates: First submitted 2017-04-30; First posted 2017-05-08 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Aortic Valve Stenosis; Valve Heart Stenosis
Keywords: aortic valve stenosis; heart valves; heart surgery
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aortic valve replacement patients: All the patients operated on aortic valve replacement in the study period at all the centers participating in the study
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: Aortic valve replacement — All surgical procedures used for both traditional and mini-invasive aortic valve replacement, as well as transcatheter valve implantation.

SUMMARY:
Traditional and transcatheter surgical treatments of severe aortic valve stenosis (SAVS) are increasing in parallel with the improved life-expectancy. Recent randomized trials (RCTs) reported comparable or non-inferior mortality with transcatheter treatments compared to traditional surgery. However, RCTs have the limitation of being a mirror of the predefined inclusion/exclusion criteria, without reflecting the "real clinical world".

Technological improvements have recently allowed the development of minimally invasive surgical accesses and the use of sutureless valves, but their impact on the clinical scenario is difficult to assess because of the monocentric design of published studies and limited sample-size. A prospective multicentre registry including all patients referred for a surgical treatment of SAVS (traditional, through full-sternotomy; minimally-invasive; or transcatheter; with both "sutured" and "sutureless" valves) will provide a "real-world" picture of available results of current surgical options, and will help to clarify the "grey zones" of current guidelines.

E-AVR is a prospective observational open registry designed to collect all data from patients admitted for SAVS, with or without coronary artery disease, in 16 cardiac surgery Centres located in six countries (France, Germany, Italy, Spain, Switzerland, and United Kingdom). Patients will be enrolled over a 2-year period and followed-up for a minimum of 5 years to a maximum of 10 years after enrolment. Outcome definitions are concordant with VARC-2 criteria and established guidelines. Primary outcome is 5-year all-cause mortality. Secondary outcomes aim at establishing "early" 30-day all-cause and cardiovascular mortality, as well as major morbidity, and "late" cardio-vascular mortality, major morbidity, structural and non-structural valve complications, quality of life and echocardiographic results.

The study protocol is approved by Local Ethics Committees. Any formal presentation or publication of data will be considered as a joint publication by the participating physician(s) and will follow the recommendations of the International Committee of Medical Journal Editors (ICMJE) for authorship.

DETAILED DESCRIPTION:
Robust early and follow-up data on the safety and efficacy of surgical TAVR, last-generation sutureless surgical valves, and minimally-invasive approaches compared with standard SAVR, with or without a contemporary (surgical or interventional) treatment of concurrent CAD, are still lacking for a real-world large population of patients at variable surgical risk. Such data is urgently required for the correct allocation of therapy in daily surgical practice. Furthermore, data on quality of life and functional echocardiographic results with different surgical alternatives might similarly help physicians in decision-making in local "Heart Teams". Data from a multicentre, real-world, open registry enrolling all patients with SAVS±CAD consecutively referred to several Centres at different European latitudes should help to answer some of these open questions.

The main strength of a prospective clinical open registry is the high external validity, given that data are collected in the settings of standard clinical practice. Moreover, large sample size enables a better estimation of event rates, and allows the investigation of hard endpoints and outcomes, by means of a wide population of patients from different institutions and with extremely limited exclusion criteria.

Importantly, clinical registries may provide data on long-term outcomes occurring after the study period of a trial. They are more practical than randomized controlled trials, require fewer resources, and have less stringent inclusion and exclusion criteria for patient enrolment. Finally, clinical findings from registries have even more significance when patient-populations derive from different geographic areas, with heterogeneous referral pathways, baseline clinical characteristics, and perioperative treatment strategies. All these features substantiate the concept of "a real world practice" underlying any "registry-study".

Therefore, the rationale of this European multicenter observational open registry is to prospectively collect data on baseline characteristics, treatment options, perioperative management and postoperative outcome of all patients consecutively undergoing surgical treatment of SAVS (regardless of gradients, AVA or AVAi)±CAD or aortic prosthetic dysfunction±CAD at 16 European university or non-university tertiary hospitals located in six European countries (France, Germany, Italy, Spain, Switzerland, and United Kingdom).

The primary aim of the study is a 5-year comparison between SAVR and surgical TAVR: we hypothesize to report a 10% superiority in terms of all-cause mortality in favor of SAVR vs TAVR. For the purpose of this study, patients will be consecutively enrolled for a 2-year period, and will be followed-up for a minimum of 5 years after the index surgical treatment. Maximum follow-up length will be 10 years after surgery.

The following surgical options will be considered:

1. SAVR with mechanical valves
2. SAVR with biological valves (either sutured or sutureless, stented or stentless)
3. Surgical TAVR (either transapical, trans-axillary, or transaortic)

Similarly, the following surgical approaches will be considered:

1. Full sternotomy
2. Mini-thoracotomy (either left-sided for TAVR or right-sided for SAVR)
3. Partial-sternotomy Patient allocation to a specific surgical procedure will be based on the local Heart Team decision at each Institution, according to standard clinical practice and current guidelines.

Patients will be recruited in a consecutive series from each institution, and their data collected in a dedicated on-line datasheet. The recruitment period will be 24 months, from 1st October 2017 to 30th September 2019. Every patient will be followed up at 30 days, 6 months, 1 year, and yearly thereafter, up to a minimum of 5 years after the index surgical procedure. Afterwards yearly follow-up will be closed at the completion of the 10th year from surgery for each patient.

On the basis of historical cohort data of local institutions, we expect to enrol a minimum of 4000 patients at the end of the first year, and a minimum of 8000 patients at the end of the second year of enrolment.

Written informed consent will be obtained from the patient or patient's authorized representative prior to enrolment in the Registry. In case of emergent surgery, informed consent will be collected from the patient's family (or legal representative) before surgery, as well as from the patient after surgery (if unable to give it before intervention). This consent will be waived in case of death or severe neurological damage precluding adequate postoperative patient informed consent. The study will be conducted in accordance with the provisions of the Declaration of Helsinki.

Data management and monitoring Data will be collected into a dedicated datasheet with predefined variables. Each patient enrolled in the Registry will be anonymized by the generation of a code consisting of the initials of the enrolling Centre (2 letters), the initial of name (1 letter) and surname (1 letter), and the date of birth (dd.mm.yyyy) (e.g. Mr. John Smith, born on February 18th, 1953; enrolled in London = LOJS18021953). It is responsibility of the E-AVR Steering Committee local member to generate the sequence to maintain anonymized the entire set of data. It is also responsibility of the E-AVR Steering Committee local member to protect confidentiality about patient identity before, during and after the trial. Accordingly, external Central Statistical Core Lab (as well as all the other E-AVR investigators) will be blinded towards patient identity.

All data will be retained in a secure location at each study-site during the conduct of the study and for the 5-years after the end of the study, when all patient identifiable paper records will be destroyed by confidential means.

Baseline characteristics, operative details and outcome data pertaining hospitalization will be prospectively collected from hospital registries. Variables and events occurring after the index hospital discharge will be collected from outpatient clinics at the individual Institutions, and linking with regional Social Security Death and Events Master files where available. In case of absent/missing data, variables and events will be collected by direct phone contact with general practitioners, and only if persistently missed by phone contact with patients and families.

Events and outcome variables will be adjudicated after agreement of two local E-AVR Investigators, and collected at local Institutions. In the event of controversy on outcome adjudication between the two local E-AVR Investigators, the outcome will be discussed and adjudicated after a final consult inside the E-AVR Steering Committee.

Storage, analysis and auditing of data will be accomplished by an independent Central Core Laboratory. Auditing of the dataset will be performed every six months by checking the data of a minimum of 40% of the patients. Data without any patient identification code will be submitted to the Principal Investigator and E-AVR Steering Committee for further data checking and merging. Incomplete or contradictory data with patient identification code will be sent from Central Core Statistical Lab to the E-AVR Steering Committee local member for further data checking, review, correction and merging. The entire set of statistical analyses will be available to all E-AVR researchers for the interpretation of data.

Ethics and Dissemination The study is approved by the local Institutional Review Boards/Ethical Committees, according to local or national guidelines for approval of registry studies. Patient's informed consent will be always obtained.

This multicenter, prospective open registry is designed with the aim of investigating a number of controversial issues regarding current treatment-options and risk factors for the surgical therapy of SAVS with or without CAD. Several studies and information are expected to derive from the data collected in the registry. These data will provide further knowledge on the mechanisms leading to adverse events during or after surgery for SAVS and help their prevention, thus allowing a "tailored" surgical approach for the treatment of this disease.

Research findings from the E-AVR registry will be disseminated among the scientific community. They will be presented at international congresses and published in peer reviewed international journals in the fields of cardiac surgery and cardiology. Any formal presentation or publication of data will be considered as a joint publication by the participating physician(s) and will follow the recommendations of the International Committee of Medical Journal Editors (ICMJE) for authorship. Data collection, analysis and writing process will be monitored by the Steering Committee of the E-AVR, which is made up of the Principal Investigator and a local Representing Member from each of the participating centres. It is expected that periodical E-AVR Steering Committee meetings will occur, every 6 months for the first 2 years, yearly thereafter up to the end of follow-up. The Members of the Steering Committee will take responsibility for the quality of data through local audit.

Investigators will be eligible for authorship if they contribute substantially to study planning, data collection, data analysis and interpretation, writing and critical review of the manuscripts. Two authors per centre will be included as main authors of each study. As a member of the Steering Committee, the local Representing Member will take any decisions on co-authorship related to his/her centre on the basis of the above criteria. Those researchers who plan a sub-study, interpret the analysis and write the article will be the first and last authors of the study. Analyses will be performed and/or monitored by an independent Central Core Statistic Laboratory. When an article is submitted to a journal with a maximum number of co-authors, the Steering Committee will decide on the authors on the basis of their contribution to the design of the study, data collection, interpretation of data, writing, and critical review of the paper.

In the event of future merging with other contemporary registries (e.g. collecting data on concurrent interventional - i.e. percutaneous transfemoral, transcarotid or trans-axillary - TAVR procedures), the co-authorship of comparative studies (e.g. between surgical and interventional treatments) will be defined by the Steering Committees of the different registries involved. However, data will not be made available for sharing until after publication of the principal results of the study. Thereafter, anonymized individual patient data will be made available for secondary research, conditional on assurance from the secondary researcher that the proposed used of the data is compliant with the MRC Policy on Data Preservation and Sharing regarding scientific quality, ethical requirements, and value for money. Anonymized data will be shared as long as the patient has agreed and consented to this. A minimum requirement with respect to scientific quality will be a publicly available pre-specified protocol describing the purpose, methods and analysis of the secondary research.

ELIGIBILITY:
Inclusion criteria

* Age >18 yy
* Isolated SAVS with or without concomitant aortic valve regurgitation
* Isolated prosthetic aortic dysfunction
* SAVS + coronary artery disease (CAD)
* Prosthetic aortic dysfunction + CAD
* Elective, urgent and emergent procedures
* Endocarditic aetiology

Exclusion criteria

* Patients undergoing concomitant mitral valve surgery, or tricuspid valve surgery, or aortic surgery (i.e. composite aortic valve and ascending aorta replacement with or without circulatory arrest), or atrial fibrillation surgery, or any other associated cardiac surgical procedure (with the exception of CABG)
* Concomitant aortic root procedure (i.e. Bentall operation, David operation, homografts, autografts)
* SAVR with techniques of aortic annular enlargement
* Porcelain aorta
* Pure aortic valve regurgitation
* Percutaneous TAVR requiring surgical cut-down (i.e. failure to comply with a full percutaneous approach, thus configuring a "hybrid procedure")
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for a surgical treatment of severe aortic valve stenosis (either traditional - through full-sternotomy - or minimally-invasive, or transcatheter - with both "sutured" and "sutureless" valves), isolated or associated with coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
5-year all-cause mortality | The outcome measure will be assessed at 5 years after surgery
  Any death occurring after surgery

SECONDARY OUTCOMES:
Follow-up all-cause mortality | The outcome measure will be assessed at time point (30 days, and yearly from 1 to 4 years after surgery, then from 6 to 10 years)
  Any death occurring after surgery
Cardiovascular mortality | The outcome measure will be assessed at time point (30 days, 1 year, and yearly up to 10 years after surgery
  Every death caused by cardiovascular events
Stroke | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Any ischemic brain injury occurring after surgery and lasting > 24 hours
Acute myocardial infarction | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Myocardial infarction (diagnosed by ECG and troponin monitoring) any time after surgery
Prolonged use of inotropes | Participants will be followed up to 72 hours after surgery
  Postoperative need for prolonged use of inotropes
Intra-aortic balloon pump | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of intra-aortic balloon pump for acute heart failure after surgery
Extra-corporeal membrane oxygenator (ECMO) | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of extracorporeal membrane oxygenation for acute heart failure after surgery
Surgical site infection | Participants will be followed up to 3 months after surgery
  Any surgical site infection occurring within three months after surgery
Blood losses | Participants will be followed 12 hours after surgery
  Amount of blood losses from drainages 12 hours after surgery
Use of blood products | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of any blood product (red blood cell, fresh frozen plasma, Octaplex, platelets) during the in-hospital stay
Nadir hematocrit | Participants will be followed up to 24 hours after the operation
  Lowest hematocrit level during the operation day
Nadir hemoglobin | Participants will be followed up to 24 hours after the operation
  Lowest hemoglobin level during the operation day
Resternotomy for bleeding | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Re-exploration for excessive bleeding
Atrial fibrillation | Participants will be followed for the duration of hospital stay (expected: 10 days)
  any new paroxysmal/permanent atrial fibrillation episode requiring or not requiring pharmacological or electrical cardioversion attempts
Cardiac conduction disturbances | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Defined as a new left bundle branch block, right bundle branch block, or atrio-ventricular block (1st, 2nd or 3rd degree).
Permanent pace-maker | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Need for new permanent pace-maker implantation
Acute kidney injury | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Severity of acute renal failure after surgery will be graded in acute kidney injury network (AKIN) stages from 1 to 3, according to Valve Academic Research Consortium (VARC)-2 criteria
Pericardial effusion | Participants will be followed up to 3 months after surgery
  Pericardial effusion requiring medical or surgical treatment
Length of stay in the intensive care unit | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Number of hours of stay in the intensive care unit after surgery
Length of in-hospital stay | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Number of days of in-hospital stay for the index procedure
Early repeat surgery | Participants will be followed up to discharge to home or to rehabilitation clinic (expected: 10 days)
  Any "redo" for failure of the index procedure before discharge to home or to rehabilitation clinic
Post procedural aortic prostheses performance | The outcome measure will be assessed at time point (30 days, 1 year and yearly thereafter up to 10 years after surgery
  A minimum set of echocardiographic data will be considered, as follows: 1) left ventricular (LV) function (EF% based on Simpson's method); 2) Indexed LV end-diastolic and end-systolic volumes and diameters;3) Wall motion score index; 4) Indexed Left atrial volume; 5) Indexed left ventricular mass; 6) native valve and prosthetic valve stenotic indexes (peak velocity, mean gradient, Doppler-velocity index, effective orifice area, indexed effective orifice area), 7) native valve and prosthetic valve regurgitation grade
Re-intervention on the aortic valve | The outcome measure will be assessed at time point (30 days, 1 year and yearly thereafter up to 10 years after surgery
  defined as any surgical or percutaneous interventional treatment that replaces (or repairs) a dysfunctional (either for structural or non-structural) aortic prosthesis implanted at the time of the index procedure.
Repeat revascularization | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Any repeat myocardial revascularization procedure performed after surgery
Aortic valve -related adverse events | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Include: 1) embolism; 2) valve thrombosis; 3) bleeding events; 3) structural valve deterioration; 4) paravalvular leakage; 5) operated valve endocarditis; 6) haemolysis
Cardioverter-defibrillator implantation | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Need for implantable cardioverter-defibrillator
Major Adverse Cardiovascular and Cerebrovascular Event (MACCE) | The outcome measure will be assessed at time point (30 days, 1 year, and yearly thereafter up to 10 years after surgery
  Defined as a composite end-point including any of the following adverse events: death from cardiovascular cause, stroke, myocardial infarction, follow-up repeated revascularization

OTHER OUTCOMES:
Quality of Life | The outcome measure will be assessed at time point (before surgery, at discharge, at 30 days, 6 months, 1 year, and yearly thereafter up to 10 years after surgery
  It will be based on eight questionnaire items reported in Short-Form 8 Health Survey questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Onorati, MD, PhD, Principal Investigator — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected into a dedicated datasheet with predefined variables. Each patient enrolled in the Registry will be anonymized by the generation of a code consisting of the initials of the enrolling Centre (2 letters), the initial of name (1 letter) and surname (1 letter), and the date of birth (dd.mm.yyyy) (e.g. Mr. John Smith, born on February 18th, 1953; enrolled in London = LOJS18021953). It is responsibility of the E-AVR Steering Committee local member to generate the sequence to maintain anonymized the entire set of data.
  Storage, analysis and auditing of data will be accomplished by an independent Central Core Laboratory. Auditing of the dataset will be performed every six months by checking the data of a minimum of 40% of the patients. Incomplete or contraddictory data with patient identification code will be sent from Central Core Statistical Lab to the E-AVR Steering Committee local member for further data checking, review, correction and merging.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from November 2019 to October 2029
Access Criteria: The overall anonimyzed datset will be shared among the participants during periodical E-AVR Steering Committee meetings. The entire set of statistical analyses derived from all the approved sub-studies will be available to all E-AVR researchers for the interpretation of data.

REFERENCES:
- [Result] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Result] Vahanian A, Baumgartner H, Bax J, Butchart E, Dion R, Filippatos G, Flachskampf F, Hall R, Iung B, Kasprzak J, Nataf P, Tornos P, Torracca L, Wenink A; Task Force on the Management of Valvular Hearth Disease of the European Society of Cardiology; ESC Committee for Practice Guidelines. Guidelines on the management of valvular heart disease: The Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology. Eur Heart J. 2007 Jan;28(2):230-68. doi: 10.1093/eurheartj/ehl428. Epub 2007 Jan 26. No abstract available. PMID 17259184
- [Result] Filsoufi F, Rahmanian PB, Castillo JG, Chikwe J, Silvay G, Adams DH. Excellent early and late outcomes of aortic valve replacement in people aged 80 and older. J Am Geriatr Soc. 2008 Feb;56(2):255-61. doi: 10.1111/j.1532-5415.2007.01535.x. Epub 2007 Nov 27. PMID 18047491
- [Result] Grossi EA, Schwartz CF, Yu PJ, Jorde UP, Crooke GA, Grau JB, Ribakove GH, Baumann FG, Ursumanno P, Culliford AT, Colvin SB, Galloway AC. High-risk aortic valve replacement: are the outcomes as bad as predicted? Ann Thorac Surg. 2008 Jan;85(1):102-6; discussion 107. doi: 10.1016/j.athoracsur.2007.05.010. PMID 18154791
- [Result] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Result] Mack MJ, Leon MB, Smith CR, Miller DC, Moses JW, Tuzcu EM, Webb JG, Douglas PS, Anderson WN, Blackstone EH, Kodali SK, Makkar RR, Fontana GP, Kapadia S, Bavaria J, Hahn RT, Thourani VH, Babaliaros V, Pichard A, Herrmann HC, Brown DL, Williams M, Akin J, Davidson MJ, Svensson LG; PARTNER 1 trial investigators. 5-year outcomes of transcatheter aortic valve replacement or surgical aortic valve replacement for high surgical risk patients with aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2477-84. doi: 10.1016/S0140-6736(15)60308-7. Epub 2015 Mar 15. PMID 25788234
- [Derived] Onorati F, Gherli R, Mariscalco G, Girdauskas E, Quintana E, Santini F, De Feo M, Sponga S, Tozzi P, Bashir M, Perrotti A, Pappalardo A, Ruggieri VG, Santarpino G, Rinaldi M, Ronaldo S, Nicolini F; E-AVR Collaborators. Outcomes comparison of different surgical strategies for the management of severe aortic valve stenosis: study protocol of a prospective multicentre European registry (E-AVR registry). BMJ Open. 2018 Feb 10;8(2):e018036. doi: 10.1136/bmjopen-2017-018036. PMID 29440154